CLINICAL TRIAL: NCT07381998
Title: The Impact of Total Thyroidectomy on Parathyroid Function and Quality of Life
Brief Title: Effects of Total Thyroid Removal on Parathyroid Function and Quality of Life
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Khalil Rafiqi, Medical Doctor, PhD student, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-155-25
Record Dates: First submitted 2026-01-21; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hypoparathyroidism Post-surgical; Quality of Life
MeSH Terms: interventions — Calcium; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- <75 % fall in intraoperative parathyroidhormone (No Intervention): Standard blood test on post operative day 1 including PTH and P-ca
- <75 % fall in intraoperative parathyroidhormone experimental (Experimental): Ommit routine blood test on post operative day 1
  Interventions: Diagnostic Test: Ommit routine blood test post operative day 1
- >75% fall in intraoperative parathyroidhormone (No Intervention): Standard treatment
- >75% fall in intraoperative parathyroidhormone experimental (Experimental): Start in Unikalk 4 times per day + d-vitamin + alfacalcidol 2 microgram 2 times per day.
  Interventions: Drug: high-dose calcium (400 mg x 4), vitamin D (19 mikg x 4), and active vitamin D supplementation (2 mikg x 2)

INTERVENTIONS:
Drug: high-dose calcium (400 mg x 4), vitamin D (19 mikg x 4), and active vitamin D supplementation (2 mikg x 2) — Standard postoperative treatment includes low-dose calcium (400 mg x 2) and vitamin D (19 mikg x 2) is initiated for all patients.
  In the intervention group, patients are randomized to standard low-dose (control group) or standard high-dose treatment including immediate postoperative initiation of high-dose calcium (400 mg x 4), vitamin D (19 mikg x 4), and active vitamin D supplementation (2 mikg x 2). In the control group, treatment with active vitamin D is only initiated in case of low PTH (<1.0 pmol/L) and low Ca2+ (<1.10 mmol/L).
  Arms: >75% fall in intraoperative parathyroidhormone experimental
Diagnostic Test: Ommit routine blood test post operative day 1 — Patients are randomized to either clinical monitoring only, without routine postoperative POD1 measurements of Ca2+ and PTH in one group or standard postoperative care, including routine blood tests for Ca2+ and PTH at POD1. All patients will have Ca2+ and PTH measured after the first postoperative week
  Arms: <75 % fall in intraoperative parathyroidhormone experimental

SUMMARY:
Postoperative hypoparathyroidism (hypoPT) is the most frequent complication after total thyroidectomy (TT). It is caused by impaired parathyroid function, leading to low calcium levels, patient discomfort, reduced quality of life (QoL), and increased healthcare costs. Traditionally, all TT patients undergo routine postoperative blood testing and standard calcium supplementation, despite varying individual risk.

This investigator-initiated project aims to improve patient outcomes by using intraoperative parathyroid hormone (ioPTH) measurements to guide postoperative care. The ioPTH decline reflect parathyroid function immediately after surgery and can identify patients at high or low risk of hypoPT.

The study is designed as a prospective, randomized controlled trial (RCT) with two arms:

Arm A (<75% ioPTH decrease): Patients randomized to either omission of routine postoperative calcium/PTH blood tests or standard monitoring.

Arm B (>75% ioPTH decrease): Patients randomized to either early high-dose calcium and vitamin D supplementation or standard therapy.

Primary outcomes are calcium and PTH levels postoperatively, incidence of hypocalcemia, and healthcare resource use. Secondary outcomes include QoL assessed by validated questionnaires (ThyPro39, SF-36, HPQ27), transient and permanent hypoPT rates, and other surgical complications.

By tailoring care to individual risk, the study aims to safely reduce unnecessary blood tests and optimize early treatment for high-risk patients. This approach has the potential to shorten hospital stays, reduce symptoms, improve QoL, and lower costs. The findings may influence clinical guidelines nationally and internationally, supporting more personalized and evidence-based management of TT patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) undergoing Total thyroidectomy with intraoperative PTH measurements.

Exclusion Criteria:

* Malabsorption (intestinal resection or gastric by-pass).
* Renal insufficiency (eGFR<30 ml/min) or deemed clinically high-risk requiring mandatory biochemical monitoring.
* Hypercalcemia (Ca2+ > 1.32 mmol/L).
* Previous thyroid or parathyroid operations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Plasma ionized calcium (Ca2+) concentration at postoperative week 1 (POD7), by POD1 biochemical testing status | 2 years
  Comparison of plasma ionized calcium (Ca2+ mmol/L) and parathyroid hormone (PTH pmol/L) after one postoperative week between patients with and without biochemical measurements at post operative day 1 (POD1.)
Plasma ionized calcium (Ca2+ mmol/L) concentration on postoperative day 2 (POD2) | 1 year
  Comparison of plasma ionized calcium (Ca2+ mmol/L) between groups at postoperative day 2 (POD2).

SECONDARY OUTCOMES:
Incidence of clinically significant hypocalcemia requiring medical intervention through 12 months | 2 years
  Proportion of participants with clinically significant hypocalcemia, defined as plasma ionized calcium (Ca2+) < 1.10 mmol/L and/or presence of symptoms of hypocalcemia, necessitating medical intervention (e.g., IV calcium and/or initiation or escalation of oral calcium ± vitamin D). Incidence will be compared between arms.
Number of postoperative blood tests through 12 months | 2 years
  Total number of postoperative blood tests per participant (count), compared between arms.
Length of index hospital stay after surgery | 2 years
  Duration of initial postoperative hospital stay per participant, measured in days (or hours), compared between arms.
Change from baseline in Thyroid-Specific Patient-Reported Outcome measure (ThyPRO-39) score through 12 months | 2 years
  Change from baseline in Thyroid-Specific Patient-Reported Outcome measure (ThyPRO-39) score assessed at baseline and at 1 week, 2 months, 6 months, and 12 months. Scores are transformed to a 0-100 scale (minimum 0, maximum 100); higher scores indicate worse thyroid-related quality of life (more symptoms/impairment).
Change from baseline in 36-Item Short Form Health Survey (SF-36) score through 12 months | 2 years
  Change from baseline in 36-Item Short Form Health Survey (SF-36) domain scores assessed at baseline and at 1 week, 2 months, 6 months, and 12 months. Each domain score ranges from 0 to 100 (minimum 0, maximum 100); higher scores indicate better health status/quality of life.
Change from baseline in Hypoparathyroidism Patient Questionnaire (HPQ-27/HPQ-28) score through 12 months | 2 years
  Change from baseline in Hypoparathyroidism Patient Questionnaire (HPQ-27/HPQ-28) score assessed at baseline and at 1 week, 2 months, 6 months, and 12 months. Scores are transformed to a 0-100 scale (minimum 0, maximum 100); higher scores indicate worse disease control / greater symptom burden
Adverse events frequency through 12 months | 2 years
  Number and proportion of participants experiencing any adverse event, compared between arms.
Incidence of transient hypoparathyroidism through 12 months | 2 years
  Proportion of participants with transient hypoparathyroidism, defined as plasma ionized calcium (Ca2+) < 1.10 mmol/L and/or need for treatment with alfacalcidol, with subsequent resolution (i.e., no longer meeting the definition and not requiring alfacalcidol) within 12 months. Incidence will be compared between arms.
Incidence of permanent hypoparathyroidism at 12 months | 2 years
  Proportion of participants meeting the hypoparathyroidism definition (plasma ionized calcium (Ca2+) < 1.10 mmol/L and/or need for alfacalcidol) that persists at 12 months, with continued need for alfacalcidol beyond 12 months. Incidence will be compared between arms.
Incidence of postoperative bleeding complication through 30 days | 2 years
  Proportion of participants with postoperative bleeding/hematoma requiring intervention (e.g., re-operation), compared between arms.
Incidence of postoperative infection through 30 days | 2 years
  Proportion of participants with postoperative infection requiring antibiotics and/or drainage, compared between arms.
Incidence of nerve injury through 12 months | 2 years
  Proportion of participants with postoperative nerve injury, defined as recurrent laryngeal nerve palsy, assessed based on patient-reported voice function and confirmed by laryngoscopy, compared between arms.
Number of resected parathyroid glands | 2 years
  Number of resected parathyroid glands per participant (count) based on pathology report, compared between arms.
Number of lymph nodes removed | 2 years
  Number of lymph nodes removed per participant (count) based on pathology report, compared between arms.
Thyroid pathology findings | 2 years
  Final thyroid pathology diagnosis based on the postoperative histopathology report, categorized as cancer, goiter, or thyrotoxicosis-related pathology, and compared between arms

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rolighed, Professor, PhD, FEBS, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No